CLINICAL TRIAL: NCT00426959
Title: Feasibility Study of Image-guided, Dynamic Dosimetry for Permanent Interstitial Prostate Brachytherapy
Brief Title: Study of Image-guided Dosimetry for Interstitial Prostate Brachytherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: J-04100
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Locally Confined Adenocarcinoma of the Prostate
Keywords: Adenocarcinoma of the prostate; PSA of less than 10 ng/mL; Combined Gleason score 6 or less; International Prostate Symptom Score (IPSS) must <or= to 18

INTERVENTIONS:
Device: Image Guided Dynamic Dosimetry — Image Guided Dynamic Dosimetry

SUMMARY:
This will be a phase I study. This phase I study is not a standard drug dose escalation study, but rather a Clinical System Performance Evaluation Trial of a therapeutic device. However for purposes of this protocol we will refer to this portion of the trial as a phase I study.

The purpose of this study is to demonstrate the feasibility and clinical practicability of the registered ultrasound and fluoroscopy (RUF) in combination with CMS Interplant system® in an initial cohort of 6 patients.

This will involve demonstrating the feasibility of using the system in an actual operating room environment as well as obtaining a preliminary assessment of the accuracy and performance of the source location algorithm by comparing with postoperative CT dosimetry.

The Primary endpoint of this study will be evaluation of the feasibility of using the RUF system and of performing real-time optimization in the operating room environment.

The Secondary endpoints of this study will be:

1. Acute and late toxicity as assessed by IPSS, SHIM, and EPIC questionnaires at multiple follow-up intervals.
2. PSA-free survival.

Study Population:

The target population will be patients with a diagnosis of adenocarcinoma of the prostate who are seen in consultation at the Johns Hopkins Hospital.

Approximately 360 patients per year with the diagnosis of prostate cancer are seen in the Department of Radiation Oncology at Johns Hopkins Hospital. Of these patients, approximately 45% have low-risk (T1a-T2a, Gleason 6 or less, PSA 10 ng/ml or less) or intermediate-risk disease and are suitable for brachytherapy based on disease risk. Within this group of patients, approximately 70% are eligible for brachytherapy based on gland size and no prior transurethral resection of prostate (TURP).

Approximately 80% of patients offered brachytherapy at consultation decide to receive their treatment at Johns Hopkins. Overall, we currently perform 2 brachytherapy procedures per week on average, for a yearly total of approximately 90 cases.

For purposes of homogeneity of treatment and patient population, this protocol will only enroll patients currently treated at this institution with brachytherapy alone, and will not enroll patients (intermediate or high risk disease) who will require external beam radiation in addition to brachytherapy.

DETAILED DESCRIPTION:
This will be a prospective Phase I study.

Subject Identification: Patient confidentiality will be maintained in accordance with Health Information Portability and Accountability Act (HIPAA) guidelines.

All participants must sign an informed consent that will describe the objectives of the study and potential risks. All patient data reported on the case reports forms will be identified by the patient's initials and study code number only.Patients shall not be identified by name. This should serve to protect the confidentiality of subjects enrolled on the trial. Clinical data and records for all subjects studied including history and physical findings, laboratory data, and results of interventions are to be maintained by the investigators in a secure, locked location. Computerized data will require password authorization(s) for access.

Description of the Recruitment Process:

Potential subjects will be identified at the time of consultation in the Department of Radiation Oncology by Dr. Song or Dr. DeWeese. If Dr. DeWeese identifies a potential patient during a consult he will refer them to Dr. Song so that Dr. Song can offer the patient the opportunity to participate. Dr. DeWeese will not offer patients the opportunity to participate but will only assist in identifying potential patients for the research team as he sees many brachytherapy cases during his consultations.

Description of the Informed Consent Process:

Only the principal investigator and those listed as co-investigators will perform the informed consent interview. The informed consent interview will take place before the patient is to be treated to ensure that the patient has adequate time to discuss the research project with family, friends, and/or other Health Care providers. During the informed consent interview the interviewer (investigator) will take as much time as needed to ensure that the potential subject understands the research project and also clearly understands that he does not have to participate in this project to receive his cancer treatment at Johns Hopkins. If the patient decides to enroll into the research project he will sign three copies of the informed consent form. One will be for his own records,one will be kept in the Clinical Research Office at Johns Hopkins, and the third one will be kept in his medical records.

Subject Assignment:

6 patients will be enrolled onto the trial. The patients will have their brachytherapy planned using a registered ultrasound and fluoroscopy (RUF) in combination with the CMS Interplant system®.

Screening Procedures for Standard Brachytherapy:

* History and physical and KPS at the time of consultation.
* Volume of the prostate based on ultrasound at the time of diagnostic biopsy. If this is not available, then patient will have prostatic volume estimated by digital rectal examination at time of consultation and confirmatory ultrasound performed in the clinic.
* Tumors are to be graded and Gleason score provided on the pathology report.
* Prostate specific antigen (PSA).
* CT scan of the pelvis. Nodes evaluated negative by imaging methods will be classified as NX.Only nodes evaluated negative by surgical sampling will be classified as N0.
* Bone scan is optional, given the low risk of positive findings in this population.
* IPSS Symptom Score at the time of consultation.

Clinical Assessments:

Once informed consent has been obtained the following assessments will be performed on the subject:

* Pre-Treatment Evaluation (to be performed within 6 weeks prior to day 1 of brachytherapy): i. History and Physical ii. IPSS, SHIM, and EPIC questionnaires (See Appendix 1 for questionnaires). iii. Serum PSA iv. Chest X-Ray v. Bone Scan (if clinically indicated) vi. CT of pelvis vii. Ultrasound volume (to be done 4 weeks to 4 days prior to day 1 of brachytherapy)
* Day 1 of Brachytherapy:

  i. Chest X-Ray> ii. CT of the Pelvis>

  > These studies can be done the day after Brachytherapy
* Day 30: 30 days (+/- 7 days) from Brachytherapy:

  i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA iv. CT of the Pelvis v. Chest X-Ray
* Month 3: 3 months (+/- 2 weeks) from Brachytherapy:

  i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA iv. Chest X-Ray
* Month 6: 6 months (+/- 4 weeks) from Brachytherapy:

  i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA
* Month 9: 9 months (+/- 4 weeks) from Brachytherapy:

  i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA
* Month 12: 12 months (+/- 4 weeks) from Brachytherapy:

  i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA
* Post 12 month follow-up patients will be followed for an additional two more years : (Note: In years 2 and 3, patients will be followed on a semiannual basis and will have the following assessments performed): i. History and Physical ii. IPSS, SHIM, EPIC questionnaires iii. Serum PSA Version 4: 07/11/2006 9

Data to be Collected:

The data that will be collected for this trial will be the results and/or findings of the procedures and assessments that are previously outlined. R

Results/findings will be abstracted from the source documents (e.g. physician notes, nursing notes, radiology reports, lab reports, etc…) and recorded onto study specific case report forms. Only medical records that have been validated by the provider will be used as source documents for data collection. The data manager assigned to this trial will be responsible for the data collection. He/She will have access to patient medical records and will record medical information from the medical record onto the case report form. The principal investigator will review the data on a monthly basis for accuracy.

Research Interventions:

RADIATION THERAPY AND RESEARCH INTERVENTIONS

The patient population who will be offered this protocol are those who are currently offered brachytherapy as standard treatment at our institution. Patients will experience no change in the procedure other than an approximately 10% increase in the duration of fluoroscopy 'on' time during the procedure. There will also be one additional CT scan post-implant to assess dosimetry at Day ~30. This is necessary to account for the effects of post-implant edema on the dosimetric parameters and source positions measurements.

Implant Volumes:

The target volume definitions are, for the most part, based upon the ICRU Report 58, Dose and Volume Specification for Reporting Interstitial Therapy.

Clinical Target Volume, CTV: Pre-implant TRUS definition of the prostate

Planning Target Volume, PTV: An enlargement of the CTV as follows:

1. Expand the TRUS definition of the prostate by 3 mm in the lateral dimension for each TRUS axial image. Thus, the lateral dimension of the prostate will increase by approximately 6 mm.
2. Expand the TRUS definition of the prostate by 3 mm in the anterior dimension for each TRUS axial image.
3. Maintain the same posterior border of the prostate as defined by TRUS.
4. Project the expanded most cephalad axial definition to a plane 3 mm cephalad to the cephalad most TRUS plane.
5. Project the expanded most caudad axial definition to a plane 3 mm caudad to the caudad most TRUS plane. The PTV is approximately 6 mm longer in the caudad-cephalad dimension than the CTV.

Evaluation Target Volume, ETV.

The ETV is defined as the post-implant CT definition of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally confined adenocarcinoma of the prostate
* PSA of less than 10 ngmL
* Combined Gleason score 6 or less, with no individual Gleason score of 4 or 5
* The patient has decided to undergo brachytherapy at the Johns Hopkins Hospital as treatment choice for his prostate cancer
* Karnofsky Performance Status greater than 70
* Prostate volume by TRUS less than 50 cc
* International Prostate symptom score must be 18 or less
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Clinical or Pathological Lymph node involvement,
* Evidence of distant metastases
* Radical surgery for carcinoma of the prostate
* Chemotherapy or pelvic radiation therapy
* Previous transurethral resection of the prostate
* Previous or concurrent cancers other than basal or squamous cell skin cancers unless disease free for at least 5 years.
* Significant obstructive symptoms
* Major medical or psychiatric illness which, in the investigator's opinion, Hip prosthesis
* Anatomic or medical condition (such as prior abdominal perineal resection or anal stricture) which would preclude the use of TRUS Implanted device or apparatus which might obstruct visibility of the implanted sources on fluoroscopy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the feasibility of using the RUF system. | 5 years
Evaluation of real-time optimization in the operating room environment. | 5 years

SECONDARY OUTCOMES:
Acute & late toxicity as assessed by IPSS, SHIM, & EPIC questionnaires. | 5 years
PSA-free survival. | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Danny Song, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at The Johns Hopkins University, Baltimore, Maryland, United States